CLINICAL TRIAL: NCT00003766
Title: Determination of Optimal O6-Benzylguanine Dose to Achieve O6-Alkylguanine-DNA Alkyltransferase Depletion in Patients With Surgically Resectable Solid Tumors
Brief Title: O6-benzylguanine Followed by Surgery in Treating Patients With Solid Tumors That Can Be Removed During Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9523; UCCRC-9523; NCI-T98-0038
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): 06-benzylguanine (100mg/m2 16 hrs before anticipated tumor tissue removal)
  Interventions: Drug: O6-benzylguanine

INTERVENTIONS:
Drug: O6-benzylguanine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of O6-benzylguanine followed by surgery in treating patients who have solid tumors that can be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the minimal O6-benzylguanine (O6-BG) dose required to deplete tumor activity to less than 10 fmol/mg protein at a specified time after administration in patients with surgically resectable solid tumors. II. Correlate tumor tissue AGT depletion with AGT depletion in peripheral blood mononuclear cells (PBMC) obtained at a specified time after O6-BG administration in these patients.

OUTLINE: This is a dose escalation study. Patients receive a single dose of O6-benzylguanine (O6-BG) IV over 1 hour at one of two dose levels. Patients undergo surgery 16-20 hours after administration of O6-BG. Up to 13 patients receive the lower dose level of O6-BG. If more than 3 patients have detectable AGT levels, additional patients receive the higher dose. The optimal biologic dose (OBD) is defined as the lowest dose level at which at least 11 of 13 patients have AGT activity less than 10 fmol/mg protein after O6-BG dosing. Patients are followed at 1 and 3 weeks post surgery.

PROJECTED ACCRUAL: A total of 13-26 patients will be accrued for this study over approximately 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed surgically resectable solid tumor

PATIENT CHARACTERISTICS: Age: Not specified Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Medically cleared for surgery No active medical or psychiatric disease that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-10; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Determine minimal dose | 2 years
  Determine minimal dose of 06-benzylguanine (06-BG) at which there is a depletion of tumor 06-BG DNA alkyltransferase activity to <10 fmol/mg protein

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Ratain, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States